CLINICAL TRIAL: NCT02097550
Title: Primary Care eHealth Intervention for Improved Outcomes in Chronic Kidney Disease
Acronym: CKD eHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-28341; 1K23DK097308-01A1 (NIH)
Record Dates: First submitted 2013-12-11; First posted 2014-03-27 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic
Keywords: Renal Insufficiency, Chronic; Kidney Failure, Chronic; Self Care; Consumer Participation; Patient Participation; Marketing; Consumer Health Information
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- eHealth Intervention (Experimental): Patients randomized to this arm will receive eHealth materials every 2-4 weeks over the 12-month intervention. However, the exact nature of timing, dose, and delivery channel will be informed by the formative research.
  Interventions: Other: eHealth Intervention
- Standard of care (No Intervention): These patients will receive the standard of care from their physician.

INTERVENTIONS:
Other: eHealth Intervention — Patients randomized to this arm will receive eHealth materials every 2-4 weeks over the 12-month intervention. However, the exact nature of timing, dose, and delivery channel will be informed by the formative research.
  Arms: eHealth Intervention

SUMMARY:
This project seeks to improve the health of patients with chronic kidney disease (CKD) by developing and testing an electronic health intervention (that will combine secure e--mail, smartphone text message, and online video materials) to promote patient use of effective medications. The information we collect on the electronic health intervention will guide future research, including a larger trial and other studies among related patient groups (e.g., racial minorities) and diseases (e.g., type 2 diabetes mellitus). The project has the potential to improve health outcomes for the millions of patients with CKD who are not yet receiving effective medications.

DETAILED DESCRIPTION:
Specific Aims:

Chronic Kidney Disease (CKD) affects over 20 million American adults. Effective medications for reducing progression remain vastly under-utilized due to well-known behavioral barriers for patients and clinicians, including the affective barriers of denial, inertia, and uncertainty. The health consequences of this poor level of medication adoption warrant development of new strategies to facilitate their use.

Moderate CKD as a Critical Juncture for Intervention: Rates of CKD are likely only to escalate as contributing conditions (e.g., type 2 diabetes, obesity) increase. With progression, patients experience costly but preventable renal and cardiovascular disease adverse outcomes (e.g., dialysis, myocardial infarction). CKD also imposes a disproportionately heavy burden on racial/ethnic minorities and those of lower socioeconomic status. There are an estimated 8 million U.S. adults with stage 3 or "moderate" CKD (defined by an estimated glomerular filtration rate (eGFR) of 30-59 mL/min/1.73m2) offering a sizeable target population for intervention. Patients with stage 3 CKD are often diagnosed at this stage of disease through routine laboratory tests performed by their primary care providers and at a time when disease progression can still be minimized. Evidence shows that use of four categories of medications (for renal protection, hypertension, diabetes, and hyperlipidemia) can slow or even halt CKD disease progression.

Underutilization of Effective Medications for CKD Exposes a Quality Gap: These effective drugs remain vastly under-utilized despite their promotion through drug formularies, practice guidelines, and clinician and patient educational campaigns, including the landmark 2002 Kidney Disease Outcomes Quality Initiative and related undertakings. National ambulatory data indicate that even among patients with CKD who are diagnosed with cardiovascular disease (CVD), only 57% are on an angiotensin converting enzyme inhibitor (ACE-I) or angiotensin receptor blocker (ARB), only 35% have achieved the target blood pressure control, and only 52% are taking a lipid-lowering agent, despite their clear benefits in high-risk populations. Those without a CVD diagnosis have comparable or even worse rates for these target measures. After a system-wide quality improvement initiative, Southern California Kaiser patients identified as having CKD still had notable quality gaps in care: though improved, 16% were missing an ACE-I/ARB, 56% had poorly controlled blood pressure, 40% had LDL over the target, and 50% of those with comorbid type 2 diabetes (diabetes) had hemoglobin A1c levels of 7% or greater.

Aim 1: Formative research-Develop the eHealth intervention Challenge: There is good evidence on how to target conscious processing for health behavior change but less on affective processing. Approach: Using a theory-based approach, we will identify the promising content, minimum dose, and delivery for an eHealth intervention to promote appropriate medication adoption. We will use observational, systematic review, and qualitative methodologies for this formative research with a special emphasis on targeting affective processing (in addition to conscious processing). Impact: We will develop an e-Health intervention that is anticipated to have an effective content, dose, and delivery.

Aim 2: Evaluative research-Pilot test the eHealth intervention in a small RCT Challenge: The eHealth intervention must be piloted and refined prior to a definitive investigation of its efficacy. Approach: We will test the eHealth intervention for feasibility in a 2-arm pilot RCT (intervention vs. usual care controls) among patients with stage 3b CKD managed in primary care and their clinicians, while also collecting data critical to designing a future efficacy trial. Randomization: patients (50/arm) will be clustered by clinician (20/arm) with targeted inclusion of 1-3/clinician. Primary outcome: 4-point "CKD score" assessing control of risk factors for CKD progression (proteinuria, blood pressure, plasma glucose, cholesterol level/calculated CVD risk). H1: the intervention group will achieve a better mean CKD score than the usual care group. Secondary outcomes: new prescriptions for the promoted medications, CKD progression, and feasibility and process data. Impact: A new intervention specifically targeted at medication adoption that is ready for evaluation in a larger efficacy RCT.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3a (eGFR 45-59) plus poorly controlled risk factors for CKD progression and/or cardiovascular disease morbidity/mortality). Our intervention is appropriate for patients with stage 3a CKD who are not yet optimized for kidney protection (in the setting of proteinuria) with ACE-inhibitors/ARBS, hypertension, diabetes and cardiovascular disease treatment. Our intervention messages promote medication classes for the optimization of these conditions and thus are appropriate for patients with stage 3a CKD who are not yet controlled for these conditions
* Stage 3b chronic kidney disease (defined as eGFR 30-44): The rationale for including patients with stage 3b CKD (defined by eGFR 30-44) but not stage 3a (eGFR 45-59) is to reduce the possibility of misclassification of those with higher eGFRs (who have little or no underlying kidney dysfunction) and to respond to evidence that patients with stage 3b CKD have much higher rates of progression to kidney failure than those with stage 3a. We chose the following inclusion criteria to optimize the balance between generalizability, participant safety, treatment adherence, and retention.
* Having a primary care provider (PCP) at UCSF, defined as an identified individual provider or provider group from whom the participant receives ongoing medical care, if needed;
* Not pregnant at study assessment.
* The ability to use a computer or smartphone
* The ability to understand English

Exclusion Criteria:

* Severe hypertriglyceridemia (TG>500 mg/dL)
* Hyperkalemia (K>5.0 mEq/L)
* Serious illness likely to preclude study completion
* Pregnancy
* Intolerance/allergy to all indicated CKD medications
* Medication management for CKD (i.e., with all of the medications/medication classes targeted for promotion by the eHealth intervention) has already been optimized
* Has never used MyChart: because MyChart use indicates a minimum level of existing familiarity with and use of eHealth materials
* Having no access to a computer or smartphone
* Plans to change primary care site.
* Family/household member of another study participant or of a study staff member;
* Already enrolled or planning to enroll in a research study that would limit full participation in this trial or confound interpretation of its results;
* Investigator discretion for clinical safety or protocol adherence reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-05; Primary Completion 2018-11-29 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
CKD metabolic control score | 12 months
  A "CKD score" will be assigned to each patient at baseline and 12-month follow-up, which will be the primary outcome of the trial. The clinical targets that comprise the CKD score consist of laboratory or clinical measurements that are routinely performed in primary care settings and, as such, are readily available in the EHR. While apparent face validity and convenience provide a good rationale for introducing the CKD score, we also recognize the need to validate the score, which we will do in stages in both Aims 1 and 2 of the study.

SECONDARY OUTCOMES:
New indicated med prescriptions | 12 months
  New prescriptions for indicated medications.
Adherence proxy measures | 12 months
  Refills for prescriptions to prescribed medications.
Patient and provider satisfaction | 12 months
  Patient and provider satisfaction will be derived from online questionnaires.
Urine albumin | 6 months
  Urine albumin
Systolic blood pressure | 6 months
  Systolic blood pressure
Hemoglobin A1c | 6 months
  Hemoglobin A1c
LDL cholesterol | 6 months
  LDL cholesterol
CKD progression | 12 months
  CKD progression measured by eGFR
Diastolic blood pressure | 12 months
  Diastolic blood pressure
HDL cholesterol | 12 months
  HDL cholesterol
Total cholesterol | 12 months
  Total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Yank, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States